CLINICAL TRIAL: NCT01008904
Title: A Pilot Phase II Trial of Magnesium Supplements to Reduce Menopausal Hot Flashes in Cancer Patients
Brief Title: Magnesium Oxide in Treating Hot Flashes in Menopausal Women With Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-12062; HM12062 (Other: VCU IRB); CDR0000650938 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-01059 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2014-02-05 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer; Cancer Survivor; Hot Flashes; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: cancer survivor; hot flashes; breast cancer; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes | interventions — Magnesium Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (magnesium oxide) (Experimental): Patients receive magnesium oxide by mouth daily or twice daily for 4 weeks.
  Interventions: Drug: magnesium oxide; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: magnesium oxide — Given PO
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
RATIONALE: Magnesium oxide may help relieve hot flashes in women with cancer.

PURPOSE: This phase II trial is studying how well magnesium oxide works in treating hot flashes in menopausal women with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if magnesium oxide supplement will decrease the frequency and severity of hot flashes by 50% in menopausal women with cancer.

Secondary

* To evaluate the effect of magnesium oxide on overall quality of life.
* To evaluate the toxicities of magnesium oxide when administered at commonly used supplement doses.

OUTLINE: Patients receive oral magnesium oxide once daily in weeks 2-5. Patients whose hot flashes are not satisfactorily controlled after 2 weeks of treatment may receive magnesium oxide twice daily in weeks 4 and 5.

Patients complete a daily hot flash diary for 5 weeks beginning 1 week before treatment. Patients also complete quality-of-life, symptom, and self-assessment questionnaires at baseline, once weekly during treatment, and at the completion of treatment.

After completion of study treatment, patients are followed up for at least 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * History of breast cancer (currently without malignant disease)
  * No history of breast cancer but wishes to avoid estrogen due to a perceived increased risk of breast cancer
* Must have bothersome hot flashes (defined by their occurrence of ≥ 14 times per week and of sufficient severity to make the patient desire therapeutic intervention) for ≥ 1 month before study entry
* Has undergone treatment for cancer (patients other than breast cancer survivors are eligible)

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Creatinine clearance ≥ 30 mL/min
* No hypersensitivity to magnesium oxide
* No medical or other condition(s) that, in the opinion of the investigator/sub-investigator, may compromise the objectives of the study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior and no concurrent antineoplastic chemotherapy, androgens, estrogens, progestational agents, or gabapentin
* More than 28 days since prior and no other concurrent investigational drugs
* Concurrent tamoxifen, raloxifene, or aromatase inhibitors allowed provided patient has been on a constant dose for > 4 weeks AND is not expected to stop the medication during the study period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-07; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Smith, MD, Principal Investigator — Massey Cancer Center

REFERENCES:
- [Result] Park H, Parker GL, Boardman CH, Morris MM, Smith TJ. A pilot phase II trial of magnesium supplements to reduce menopausal hot flashes in breast cancer patients. Support Care Cancer. 2011 Jun;19(6):859-63. doi: 10.1007/s00520-011-1099-7. Epub 2011 Jan 27. PMID 21271347

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled female patients with bothersome hot flashes (defined by their occurrence ≥14 times per week and of sufficient severity to make the patient desire therapeutic intervention for ≥ 1 month prior to study entry) after undergoing treatment for cancer. Patients were recruited from the Massey Cancer Center oncology clinics.
Pre-assignment Details: Of the 31 patients enrolled, 29 received treatment. 25 completed treatment and were analyzed.
Period: Overall Study
Arm/Group | Supportive Care (Magnesium Oxide)
Started | 29
Completed | 25
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 2
Not completed — unexpected unrelated surgery | 1

BASELINE CHARACTERISTICS:
Population: patient who started study treatment
Groups:
- Supportive Care (Magnesium Oxide): Patients receive magnesium oxide PO QD or BID for 4 weeks.
Arm/Group | Supportive Care (Magnesium Oxide)
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Percent Difference in Hot Flash Activity (Score) Between Baseline and End of Treatment (Week 5)
Description: Hot flash score (frequency x severity) at baseline was compared to the end of treatment. The number of flashes in a 24 hour day and a score combining the number and severity of hot flashes (ie, 1 point for mild, 2 points for moderate, 3 points for severe and 4 points for very severe.
Time Frame: from baseline to week 5
Population: 25 patients completed the complete study and were analyzed
Measure: Mean (Standard Error); unit: percentage of difference
Arm/Group | Supportive Care (Magnesium Oxide)
Number analyzed (Participants) | 25
percentage of difference | -50.4 (40.9)

2. Secondary Outcome: Difference in Quality of Life
Description: Mayo Clinic Uniscale instrument (6 questions with each question rating 0=as bad as it can be and 10=as good as it can be). A lower score is considered to be a better outcome.
Time Frame: from baseline to week 5
Population: Participants who completed treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Supportive Care (Magnesium Oxide)
Number analyzed (Participants) | 25
units on a scale | 0.14 (0.3)

ADVERSE EVENTS:
Time Frame: Study start to study completion. (5 weeks
Arm/Group | Supportive Care (Magnesium Oxide)
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 2/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Magnesium Oxide) (N=29)
Surgery (Skin and subcutaneous tissue disorders) | 1 (1) — unrelated due to seroma involving the left breast flap, after bilateral TRAM flap
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Magnesium Oxide) (N=29)
Diarrhea (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No